CLINICAL TRIAL: NCT03368469
Title: A Pilot Study of the Tolerability and Efficacy of Transcranial Direct Current Stimulation (tDCS) in Children and Adolescents With Epilepsy and Comorbid Depression
Brief Title: Transcranial Direct Current Stimulation (tDCS) in Children and Adolescents With Epilepsy and Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study team was unable to recruit and enroll subjects. The study is now closed.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul E. Croarkin, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-001007
Record Dates: First submitted 2017-12-01; First posted 2017-12-11 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Depressive Disorder; Generalized Epilepsy
Keywords: Transcranial; Stimulation
MeSH Terms: conditions — Depressive Disorder; Epilepsy, Generalized | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- transcranial direct current stimulation (Experimental): Transcranial direct current stimulation (35 sq cm anode over left dorsolateral prefrontal cortex, 35 sq cm cathode over right supraorbital area, 1 mA current, 20 min per treatment session, 1 session per day, 10 treatment sessions over two weeks)
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — The Soterix Medical 1×1 Low Intensity Transcranial DC Stimulator Model 1300A is an investigational device manufactured by Soterix Medical, Inc. (New York, NY, USA). It is designed for use in noninvasive transcranial stimulation of the brain by delivering low-intensity electrical current to the scalp through two electrodes.
  Other Names: Soterix Medical Model 1300A

SUMMARY:
The proposed study seeks to obtain preliminary signal of the tolerability and efficacy of transcranial direct current stimulation (tDCS) for depressive symptoms in a sample of adolescents with depression and epilepsy. Additionally, effects of tDCS will be assessed via electroencephalographic, cognitive, and psychosocial measures.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) has been investigated extensively in recent years for the treatment of depression. Meta-analysis of individual patient data indicates that tDCS results in improvement in depressive symptoms, with efficacy comparable to antidepressant medications and repetitive transcranial magnetic stimulation (rTMS), while tDCS offers advantages over other treatments, including side effect profile, cost, and portability. tDCS has been employed to a more limited extent in children and adolescents for psychiatric conditions other than depression, as well as in both adults and children with epilepsy, with excellent tolerability and a mild adverse effect profile. The proposed protocol aims to extend the use of tDCS for treatment of depression in children with epilepsy (CWE), a population with a very high prevalence of depression and a significant need for additional treatment options, particularly nonpharmacologic treatments, due to challenges with the use of antidepressant medications and other non-invasive brain stimulation (NIBS) techniques in CWE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized epilepsy (confirmed by neurologist)
* Diagnosis of depressive disorder (confirmed by psychiatrist), with CDRS-R score ≥ 40
* Parent/guardian ability to provide written informed consent in English, with child/adolescent participant able to provide assent (for participants <18 years of age), or participant ability to provide written informed consent in English (for participants ≥18 years of age)
* Antidepressant medications (SSRI or SNRI) permitted, provided that no dosing change has occurred in two months prior to baseline assessments; antidepressant medication not required for enrollment
* AED medications (with exceptions listed below in exclusion criteria) permitted, provided that no change in AED regimen has occurred in two months prior to baseline assessments (except for weight/growth-related dosing changes); AED not required for enrollment

Exclusion Criteria:

* Presence of pacemaker or metallic implant (with the exception of orthodontic hardware)
* Prior surgical intervention for epilepsy
* More than one generalized tonic-clonic (GTC) seizure during two months prior to enrollment
* AED regimen change during two months prior to baseline assessments (except dosing adjustments made strictly due to growth/weight change)
* Antidepressant medication change during two months prior to baseline assessments
* Lifetime history of manic/hypomanic episode or psychotic disorder
* Autism spectrum disorder (ASD) diagnosis
* Documented history of intellectual disability (documented full-scale IQ greater than two standard deviations below mean)
* Current or recent (two months prior to baseline assessments) active substance use disorder
* Imminent risk of suicide or medically serious self-injurious behavior (as evaluated by board-certified child and adolescent psychiatrist)
* Current pregnancy or positive urine pregnancy test
* Prohibited concomitant medications include: regularly scheduled benzodiazepines (except clobazam); barbiturates; neuroleptic/antipsychotic medications; lithium.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Children's Depression Rating Scale - Revised (CDRS-R) total score | 2 weeks
  clinician-rated continuous measure of depression severity based on participant and parent interviews

SECONDARY OUTCOMES:
Children's Depression Rating Scale - Revised (CDRS-R) total score | 3 months, 6 months
  clinician-rated continuous measure of depression severity based on participant and parent interviews
Quick Inventory of Depressive Symptoms - Adolescent - Self-Report (QIDS-A17-SR) total score | day 1, day 5, day 10, 3 months, 6 months
  participant-reported continuous measure of depression severity
tDCS Adverse Effects Survey | days 1-10, 2 weeks, 3 months, 6 months
  standardized self-report questionnaire for active reporting of adverse effects; will be used to calculate incidence of all adverse effects (AEs) and severe adverse effects (SAEs) as well as incidence of specific AEs/SAEs
Columbia Suicide Severity Rating Scale (C-SSRS) | day 1, day 5, day 10, 2 weeks, 3 months, 6 months
  measure of suicidal ideation and behavior based on clinician interview
Young Mania Rating Scale (YMRS) | day 5, 2 weeks
  measure of manic symptoms based on clinician interview/observation
Affective Reactivity Index (ARI) | 2 weeks, 3 months, 6 months
  parent- and participant-report questionnaires regarding symptoms of irritability
Mayo Seizure Frequency Assessment | 2 weeks, 3 months, 6 months
  parent- and participant-report questionnaires regarding seizure frequency
Liverpool Seizure Severity Scale (1998 revision) | 2 weeks, 3 months, 6 months
  parent-/participant-report questionnaire regarding seizure severity and quality
Impact of Pediatric Epilepsy Scale (IPES) | 2 weeks, 3 months, 6 months
  parent-report questionnaire regarding impact of epilepsy of quality of life
Quality of Life in Epilepsy Inventory for Adolescents (QOLIE-AD-48) | 2 weeks, 3 months, 6 months
  participant-report questionnaire regarding impact of epilepsy of quality of life
NIH Toolbox® for Assessment of Neurological and Behavioral Function | 2 weeks
  validated and age-normed computer-administered battery of measures assessing cognitive functioning
Electroencephalography (EEG) | 2 weeks
  objective electrophysiologic data on brain activity; a board-certified epileptologist will manually quantify the maximal number of spike-wave discharges per 20-second recording, the longest run of epileptiform discharges, and, if sleep EEG is obtained, the spike-wave index; additionally, broadband EEG will be obtained to assess indices of cortical excitability, such as relationships between slow oscillations, interictal epileptiform discharges, and sleep architecture

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Croarkin, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Lee JC, Lewis CP, Daskalakis ZJ, Croarkin PE. Transcranial Direct Current Stimulation: Considerations for Research in Adolescent Depression. Front Psychiatry. 2017 Jun 7;8:91. doi: 10.3389/fpsyt.2017.00091. eCollection 2017. PMID 28638351
- [Background] Hameed MQ, Dhamne SC, Gersner R, Kaye HL, Oberman LM, Pascual-Leone A, Rotenberg A. Transcranial Magnetic and Direct Current Stimulation in Children. Curr Neurol Neurosci Rep. 2017 Feb;17(2):11. doi: 10.1007/s11910-017-0719-0. PMID 28229395
- [Background] Muszkat D, Polanczyk GV, Dias TG, Brunoni AR. Transcranial Direct Current Stimulation in Child and Adolescent Psychiatry. J Child Adolesc Psychopharmacol. 2016 Sep;26(7):590-7. doi: 10.1089/cap.2015.0172. Epub 2016 Mar 30. PMID 27027666
- [Background] Godinho MM, Junqueira DR, Castro ML, Loke Y, Golder S, Neto HP. Safety of transcranial direct current stimulation: Evidence based update 2016. Brain Stimul. 2017 Sep-Oct;10(5):983-985. doi: 10.1016/j.brs.2017.07.001. Epub 2017 Jul 8. No abstract available. PMID 28751225
- [Background] Krishnan C, Santos L, Peterson MD, Ehinger M. Safety of noninvasive brain stimulation in children and adolescents. Brain Stimul. 2015 Jan-Feb;8(1):76-87. doi: 10.1016/j.brs.2014.10.012. Epub 2014 Oct 28. PMID 25499471
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials